CLINICAL TRIAL: NCT00855101
Title: An Open-Label, Intravenous (6/4 Mg/Kg Q12h) To Oral Switch (200 Mg Q12h), Multiple Dose Study To Evaluate The Pharmacokinetics, Safety And Tolerability Of Voriconazole In Healthy Male And Female Adults
Brief Title: A Pharmacokinetic And Safety Study Of Voriconazole In Healthy Male And Female Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A1501092
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics and safety of voriconazole intravenous oral adults
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- voriconazole (Experimental)
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — 6 mg/kg IV q12h on Day 1, and 4 mg/kg IV q12h on Days 2-7, then switch to 200 mg oral tablet q12h on Days 8-14.
  Other Names: Vfend

SUMMARY:
This study is to assess the plasma concentration-time profile of voriconazole in adults receiving 7-day intravenous treatment and 6.5-day oral treatment. This study is also to assess the safety profile of voriconazole during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects from 18 and 55 years old.
* Body weight between 40 kg (88 lbs) and 100 kg (220 lbs).

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, ocular, neurologic, or allergic disease.
* Subjects with any condition possibly affecting drug absorption, eg, gastrectomy.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetics of voriconazole following an intravenous to oral switch regimen in healthy adults | 14 days

SECONDARY OUTCOMES:
The safety and tolerability of voriconazole following an intravenous to oral switch regimen in healthy adults | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501092&StudyName=A%20Pharmacokinetic%20And%20Safety%20Study%20Of%20Voriconazole%20In%20Healthy%20Male%20And%20Female%20Adults